CLINICAL TRIAL: NCT02762175
Title: 3D Volumetric Changes in the Upper Airway After Maxillomandibular Advancement in Obstructive Sleep Apnea Syndrome Patients and the Implication on Quality of Life: A Prospective Registry
Brief Title: 3D Volumetric Changes in the Upper Airway After MMA in OSAS Patients and the Implication on QOL: A Prospective Registry
Acronym: MMA-OSAS
Status: Recruiting | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Nathalie Neyt, maxillofacial surgeon, AZ Sint-Jan AV
Other Study IDs: B049201627590
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: maxillomandibular advancement; obstructive sleep apnea; apnea-hypopnea index; quality of life
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background

Obstructive sleep apnea syndrome (OSAS) is a sleep-related breathing disorder characterized by intense snoring and repetitive complete or partial obstructions of the upper airway during sleep together with daytime sleepiness. Several non-invasive therapeutical options exist, however, they do not offer a permanent improvement. Maxillomandibular advancement (MMA) surgery is a procedure which changes the upper airway in a permanent way.

Objectives

The investigators aim to develop a prospective database registering 3D volumetric changes of the upper airway and its anatomic subregions, the apnea-hypopnea index (AHI) and quality of life (QOL) of all consecutive patients eligible for MMA, performed by Dr. Neyt. Patient demographics, detailed virtual cone-beam computed tomography (CBCT) planning parameters, orthognathic surgery, polysomnographic and QOL data are being collected during consecutive visits within the framework of routine practice.

Design

A prospective, observational cohort study

Study center

General Hospital (AZ) Sint-Jan Brugge-Oostende

Population

The investigators would like to include all OSAS patients (AHI ≥ 5) requiring a MMA by Dr. Neyt starting from January 2015.

Endpoints

The investigators aim to collect data that could provide information about the advantages and disadvantages of the routinely performed 3D CBCT preoperative MMA surgery planning for OSAS patients, regarding 3D volumetric changes of the upper airway and its anatomic subregions and quality of life (QOL) in a subjective manner with the Epworth Sleepiness Scale (ESS) and the OSAS questionnaire and in an objective manner with evaluation of the apnea-hypopnea index (AHI).

Duration

In light of the continuous improvement of patient care, a database will be maintained from January 2015 onwards to enable registration of large-scale OSAS patient data.

Conclusions

Development of a database registering 3D CBCT planning, polysomnographic data and quality of life (QOL) of all consecutive patients eligible for MMA, will provide more information about potential patient, virtual planning and surgical factors influencing accuracy of MMA, and the associated biological benefits of this procedure on the upper airway volume, the AHI and general QOL. Moreover, registration of those results could function as a measurement of quality of care, or could be used for sample size calculation for future large multicenter prospective trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages
* Patients of all genders
* Patients diagnosed with OSAS, based on an AHI ≥ 5
* All consecutive OSAS patients operated by N. Neyt from January 2015 onwards

Exclusion Criteria:

* Patients not eligible according to abovementioned criteria
* Patients with morbid obesity (BMI >35), if judged non-eligible by the treating surgeon

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all OSAS patients (AHI ≥ 5) requiring a MMA by Dr. Neyt starting from January 2015
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
postoperative apnea-hypopnea index, measured with polysomnography | 6-12 months

SECONDARY OUTCOMES:
3D volumetric changes of the upper airway, measured with cone-beam CT | 4-6 months
quality of life, measured with epworth sleepiness scale | 4-12 months
quality of life, measured with OSAS questionnaire | 4-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Neyt, MD, Principal Investigator — Division of Maxillofacial Surgery, Department of Surgery, AZ Sint-Jan Brugge-Oostende AV
Locations (1):
- Division of Maxillofacial Surgery, Department of Surgery, AZ Sint-Jan Brugge Oostende AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No